CLINICAL TRIAL: NCT06363162
Title: Evaluate the Effectiveness and Safety of the Raman IVD Analyzer in the Molecular Diagnosis of Gliomas During Surgery, Using Samples From Brain Resection Tissue (Ambispective, Multicenter, Blind Evaluation, Single Group Target Value Method)
Brief Title: Evaluate the Effectiveness and Safety of Raman IVD Analyzer in the Molecular Diagnosis of Gliomas During Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: West China Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Capital Medical University (Other); Jiangsu Raman Medical Equipment Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LRR202404
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Glioma
Keywords: Molecular subtype; Raman; intraoperative; surgery
MeSH Terms: conditions — Glioma | interventions — Immunohistochemistry; Genetic Testing

STUDY DESIGN:
Intervention Model Description: The same sample was diagnosed using Raman spectroscopy and immunohistochemistry or genetic test, respectively. Calculate the AUC, the accuracy, the sensitivity and specificity of a Raman analyzer using immunohistochemistry or genetic test results as the gold standard.
Masking Description: Blind assessment: Researchers using Raman analyzer during surgery are not aware of the subjects' preoperative diagnostic results, while researchers conducting immunohistochemistry or genetic test after surgery are not aware of the subjects' preoperative diagnostic results and the diagnostic results of Raman analyzer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perform two different tests on the same sample (Experimental): Perform the diagnosis of Raman analyzer and immunohistochemistry or genetic test on the same sample.
  Interventions: Diagnostic Test: Immunohistochemistry or genetic test

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry or genetic test — Perform two diagnostic methods on the same sample
  Other Names: Raman analyzer diagnosis

SUMMARY:
To distinguish various molecular subtypes of gliomas by spectra data obtained from Raman analyzer, including IDH mutant, 1p/19q-codeleted, ATRX deletion, TERT promoter mutation, MGMT promoter methylation, EGFR amplification, H3 K27-altered, TP53 mutant, PTEN deficiency, ki 67, AQP4, VEGF, and so on, comparing with the results of Immunohistochemistry or genetic test on the same brain tissue samples.

DETAILED DESCRIPTION:
1500 samples were included retrospectively with the spectra data obtained from Raman analyzer to establish clinical intelligence model, modifying the analyzer. Based on statistical calculations, 200 glioma samples will be included in the trial in all trial centers prospectively. Compare the results between the Raman analyzer and Immunohistochemistry or genetic test results. And calculate the AUC, the accuracy, sensitivity, the specificity, and other indicators of Raman analyzer.

During surgery, core tissue samples were taken from subjects. The test samples size:0.2cm<length diameter ≤ 2cm. The sample testing result is based on the Raman test points. Then take the same tissue sample for Immunohistochemistry or genetic test.

Statistical description of all data, including baseline data, all efficacy indicators, and all safety data. The measurement data give the mean, standard deviation, minimum, maximum, median,25 quantile and 75 quantile; Provide frequency and composition ratio for counting data. The baseline data was analyzed using the Full Analysis Set (FAS); The effectiveness analysis adopts FAS and PPS; The security analysis uses the Security Dataset (SS).

ELIGIBILITY:
Inclusion Criteria:

* Patients who plan to undergo brain lesion tissue resection surgery or have preoperative clinical diagnosis of gliomas and plan to undergo biopsy;
* Patients with clinical diagnosis of initial solitary gliomas, or initial solitary intracranial masses or initial non occupying lesions that do not exclude gliomas (such as intracranial metastatic lesions, intracranial infectious lesions, intracranial demyelinating lesions, central nervous system lymphoma, etc.), who have not received radiotherapy or chemotherapy in the past based on their medical history;
* The patient or their guardian can understand the research purpose, demonstrate sufficient compliance with the trial protocol, consent for immunohistochemistry or genetic test, and sign an informed consent form;
* It is possible to obtain tissue samples with a length diameter greater than 0.2cm. Patients diagnosed with initial solitary glioma should take core or marginal tissue, while patients diagnosed with initial single intracranial mass or initial non mass lesions but maybe with gliomas should be taken core tissue.

Exclusion Criteria:

Investigator judge that it is not suitable for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve | Through study completion, an average of 1 year
  The Area Under the Curve of the ROC curve illustrates the performance of Raman analyzer for the diagnosis of molecular subtype in glioma, confirmed by immunohistochemistry or genetic test.
Accuracy | Through study completion, an average of 1 year
  The proportion of tissue samples with consistent results between Raman analyzer detection and immunohistochemistry or genetic test.

SECONDARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  Among one kind of molecular subtype samples determined by immunohistochemistry or genetic test, the percentage of samples detected by Raman analyzer as the same molecular subtype.
Specificity | Through study completion, an average of 1 year
  Among one kind of molecular subtype samples determined by immunohistochemistry or genetic test, the percentage of samples detected by Raman analyzer as the different molecular subtype.
Kappa coefficient | Through study completion, an average of 1 year
  Kappa coefficient≥0.75 indicates high consistency; 0.75>Kappa coefficient≥0.4, considered consistent; If the Kappa coefficient is less than 0.4, it is considered inconsistent.
Time consumption for the Raman analyzer in detection | Through study completion, an average of 1 year
  Time required from emitting laser to completing single point detection
Adverse Event Incidence Rate | During the surgery
  Number of subjects with AE/total number of subjects ×100%
Serious Adverse Event Incidence Rate | During the surgery
  Number of subjects with SAE/total number of subjects ×100%
Operator adverse events | Through study completion, an average of 1 year
  Possible damage to device operators during the use and maintenance of the Raman analyzers

CONTACTS AND LOCATIONS:
Overall Officials: Qing Mao, Principal Investigator — West China Hospital; Dongming Yan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Shouwei Li, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China